CLINICAL TRIAL: NCT06567106
Title: Investigation of Cardiac Function Following Low-Intensity Ultrasound Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ShanghaiTech University (Other)
Responsible Party: Principal Investigator, Bingbing Cheng, Assistant Professor, ShanghaiTech University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Q2024-004
Record Dates: First submitted 2024-08-14; First posted 2024-08-22 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Cardiac Function
Keywords: Ultrasound; Heart; Cardiac function

STUDY DESIGN:
Intervention Model Description: Each participant is randomly assigned to receive either ultrasound intervention at varying intensities or sham control.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and outcomes assessors are blinded to the experimental condition.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Ultrasound application at minimal intensity (Experimental): Apply minimal-intensity ultrasound to the participant. The intensity is below 2 W/cm².
  Interventions: Other: Ultrasound application
- Ultrasound application at mild intensity (Experimental): Apply mild-intensity ultrasound to the participant. The intensity is below 3 W/cm².
  Interventions: Other: Ultrasound application
- Ultrasound application at medium intensity (Sham Comparator): Apply medium-intensity ultrasound to the participant. The intensity is below 5 W/cm².
  Interventions: Other: Ultrasound application
- No ultrasound application (Sham Comparator): No ultrasound application to the participant.
  Interventions: Other: No ultrasound application

INTERVENTIONS:
Other: Ultrasound application — Apply ultrasound to the participant within a safe range.
  Arms: Ultrasound application at medium intensity; Ultrasound application at mild intensity; Ultrasound application at minimal intensity
Other: No ultrasound application — No ultrasound application to the participant.
  Arms: No ultrasound application

SUMMARY:
The goal of this clinical trial is to investigate the influence of ultrasound on cardiac functrion.

The main question it aims to answer is:

How will ultrasound affect the cardiac function?

Researchers will： Apply ultrasound to the body and observe cardiac functions.

Participants will:

Receive ultrasound application and physiological signal monitoring.

DETAILED DESCRIPTION:
All procedures conducted in this trial comply with the ethical standards of the relevant national and institutional committees on human experimentation and with the Helsinki Declaration of 1975, as revised in 2008. All procedures were approved by the Research Ethics Committee of ShanghaiTech University (Q2024-004).

The primary outcome is heart rhythm. It will be measured by electrocardiogram. The secondary primary outcome is the incidence of treatment-related adverse events. It will be measured by electrocardiogram and observation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals without significant diseases or chronic conditions.
* Aged between 18 and 65 years.
* Voluntary participation with signed informed consent.
* No history of cardiovascular disease.

Exclusion Criteria:

* Individuals with heart disease or other conditions that may affect cardiac function measurement.
* Individuals with implanted electronic devices such as pacemakers or defibrillators.
* Those on medications that significantly alter heart rate, such as beta-blockers, unless under stable control for a specific period.
* Individuals at risk of severe complications.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2027-10-10 (Estimated); Study Completion 2027-10-10 (Estimated)

PRIMARY OUTCOMES:
Heart rhythm. | Throughout the intervention, an average of 1 hour.
  Monitor participants' electrocardiogram before, during and after ultrasound application. Calculate heart rate from the electrocardiogram signal. The change of heart rate is calculated as the rate of change relative to the baseline heart rate. Aggregate the data and do statistical analysis. Data will be presented as mean with standard deviations.
Incidence of treatment-related adverse events. | Baseline, during the intervention (an average of 1 hour) and immediately after the intervention (same day, approximately 1 hour after baseline).
  The incidence of treatment-related adverse events includes both minor (such as localized discomfort, transient arrhythmias, mild chest pain, short-term dizziness, nausea, and temporary shortness of breath) and severe adverse events (including sustained arrhythmias, new-onset heart failure, significant myocardial injury, embolic events, or death).

CONTACTS AND LOCATIONS:
Locations (1):
- Bingbing Cheng, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-10-10): https://cdn.clinicaltrials.gov/large-docs/06/NCT06567106/Prot_SAP_ICF_001.pdf